CLINICAL TRIAL: NCT03541356
Title: A Phase IIa, Randomized, Double Blind, Placebo Controlled, Single Ascending Dose, Safety and Pharmacokinetic/Pharmacodynamic Study of INP103 (POD L-dopa) Administered in the Presence of DCI to L-dopa Responsive Parkinson's Disease Patients
Brief Title: Therapeutic Potential for Intranasal Levodopa in Parkinson's Disease -Off Reversal
Acronym: THOR201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Impel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INP103-201
Record Dates: First submitted 2018-04-05; First posted 2018-05-30 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinsons; L-dopa; levodopa; ON; OFF; PD; POD device; I231; benserazide; Precision olfactory delivery; MDS-UPDRS; Carbidopa; DCI; Decarboxylase Inhibitor
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Carbidopa

STUDY DESIGN:
Intervention Model Description: Thirty-Two (32) to Thirty-Six (36) subjects will be randomized to treatment or placebo. INP103 is a drug-device combination product containing a drug component, L-dopa, and device component, the I231 Precision Olfactory Delivery (POD) device. In Cohorts 1, 2, and 3, L-dopa will be administered intranasally in single doses of one (35 mg), two (70 mg) or four (140 mg) puffs of INP103, 60 minutes after oral benserazide hydrochloride 25 mg.
  In Cohort 4 the INP103 formulation will contain L-dopa:carbidopa administered nasally. Dosing will take place once OFF episode is confirmed and will not include predosing with oral benserazide.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo
- L-dopa 35 mg (Active Comparator)
  Interventions: Combination Product: L-dopa 35 mg
- L-dopa 70 mg (Active Comparator)
  Interventions: Combination Product: L-dopa 70mg
- L-dopa 140 mg (Active Comparator)
  Interventions: Combination Product: L-dopa 140 mg
- L-dopa 70 mg/carbidopa 7 mg (Active Comparator)
  Interventions: Combination Product: L-dopa 70mg/carbidopa 7mg

INTERVENTIONS:
Combination Product: Placebo — Delivered via the I231 POD (Precision Olfactory Delivery) device
  Arms: Placebo
Combination Product: L-dopa 35 mg — Delivered via the I231 POD (Precision Olfactory Delivery) device via one puff to one nostril
  Arms: L-dopa 35 mg
Combination Product: L-dopa 70mg — Delivered via the I231 POD (Precision Olfactory Delivery) device with two puffs, one to each nostril
  Arms: L-dopa 70 mg
Combination Product: L-dopa 140 mg — Delivered via the I231 POD (Precision Olfactory Delivery) device with four puffs, two to each nostril
  Arms: L-dopa 140 mg
Combination Product: L-dopa 70mg/carbidopa 7mg — Delivered via the I231 POD (Precision Olfactory Delivery) device with two puffs, one to each nostril
  Arms: L-dopa 70 mg/carbidopa 7 mg

SUMMARY:
A Phase IIa, Randomized, Double Blind, Placebo Controlled, Single Dose, Safety and Pharmacokinetic/Pharmacodynamic Study of INP103 (POD L-dopa) Administered in the Presence of Decarboxylase Inhibitor to L-dopa Responsive Parkinson's Disease Patients

DETAILED DESCRIPTION:
This is a Phase IIa randomized, double-blind, placebo-controlled, single dose study to compare the safety, tolerability and PK/PDyn of intranasal L-dopa following administration of INP103 in the presence of L-dopa decarboxylase inhibitor (DCI) during an OFF episode.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females, 40 to 80 years of age (inclusive) at the time of Screening (Visit1)
2. Diagnosed with Idiopathic PD (by UK Brain Bank Criteria) with Modified Hoehn & Yahr (H&Y) Stage I-III during an ON period at Visit 1
3. Subjects who are prone to (and recognize) OFF episodes (when their usual PD medication has worn off)
4. Shown to be responsive to L-dopa medication (≥ 30% improvement in MDS-UPDRS Part III Motor Examination score) as assessed during the Screening period (Visit 2)
5. On a stable dose of L-dopa containing medication for at least 2 weeks prior to Visit 1 (up to 1200 mg/day) with no single dose exceeding 250 mg. All other anti-PD medication (e.g. dopamine agonists [DAs], monoamine oxidase-B inhibitor (MAOB-I) or catechol-O-methyl transferase (COMT) inhibitors ARE allowed if the subject has been on a stable dose for at least 30 days prior to Visit 1.
6. Willing to omit their (usual) PD drugs (e.g. usual regular anti-PD medication including any L-dopa containing medication, DAs and/or COMT inhibitors and any required anti-OFF treatment) from 22:00 pm the evening prior to study dosing until 120 minutes post study treatment dosing.

   Cohorts 1, 2 and 3 ONLY WILL take oral benserazide 25 mg on arrival at the research site (at 60 ± 5 minutes before dosing with INP103 or placebo).

   Cohort 4 will omit oral benserazide and subjects may be dosed once OFF episode has been confirmed and all baseline assessments have been completed.
7. If female and of childbearing potential must agree to use adequate contraception (see Section 4.4) during the study
8. Able and willing to attend the necessary visits at the study centre
9. Willing to provide voluntary written informed consent signed prior to entry into the study

Exclusion Criteria:

1. Severe dyskinesia (defined as per MDS-UPDRS) during a 'normal day' that would significantly interfere with the subject's ability to perform study assessments
2. In receipt of L-dopa containing medication at > 1200 mg/day
3. History of significant psychotic episode(s) within the previous 12 months in the opinion of the Investigator, or currently receiving anti-psychotic medication at a moderate dose (quetiapine >50 mg/day, risperidone >1 mg/day or olanzapine >2.5 mg/day)
4. Mini Mental State Examination (MMSE) ≤ 25 as documented within the previous 36 months or as assessed by Investigator during Screening
5. History of suicidal ideation or attempted suicide within previous 12 months
6. Narrow-angle glaucoma
7. Presence of skin lesions that, in the opinion of the Investigator, may be cancerous
8. Females who are pregnant, planning a pregnancy or lactating
9. Subjects with any underlying physical condition that, in the opinion of the Investigator, would make it unlikely that the subject will comply with or be able to complete the study requirements
10. Use of any medication likely to interact with benserazide, carbidopa or INP103 (see Appendix 5)
11. Laboratory test abnormalities at Screening (Visit 1) deemed clinically significant by the Investigator.
12. History or presence of alcoholism or drug abuse within the 2 years prior to INP103 or placebo dosing
13. Administration of an investigational product in another trial within 30 days or 5 half-lives (whichever is longer) prior to INP103 or placebo dosing
14. Significant nasal congestion, physical blockage in either nostril, or significantly deviated nasal septum as evaluated by the PI or other suitably trained healthcare professional
15. Subjects who have previously shown hypersensitivity to L-dopa or benserazide (for Cohorts 1, 2 and 3), or L-dopa or carbidopa (for Cohort 4) or any of their excipients

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Shrewsbury, MD, Study Chair — Impel NeuroPharma, Seattle, WA (USA); Terry O'Brien, MD/Prof, Principal Investigator — The Alfred Hospital, Melbourne, VIC (AUS)
Locations (5):
- Australia (5):
  - The Brain and Mind Centre / Scientia Clinical Research, Sydney, New South Wales
  - Q-Pharm, Brisbane, Queensland
  - The Mater Hospital, Brisbane, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - Perron Institute, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parkinson's disease patients at movement disorder clinics in Australia
Pre-assignment Details: Confirmation of L-dopa responsiveness at Visit 2, prior to randomization
Period: Overall Study
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Started | 8 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 1 | 3 | 5 | 18
  >=65 years | 2 | 3 | 5 | 3 | 1 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 3 | 12
  Male | 5 | 4 | 4 | 4 | 3 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 6 | 6 | 6 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 4 | 6 | 6 | 6 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 8 | 6 | 6 | 6 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Assessment of treatment emergent adverse events after single dosing with INP103 (L-dopa or L-dopa/carbidopa)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participants | 5 | 5 | 3 | 4 | 5

2. Secondary Outcome: AUC0-2hr for L-dopa
Description: Area under the Plasma Concentration-time Curve for L-dopa from Time = 0 to Time = 2 hours post dose. For the L-dopa 35 mg, L-dopa 70 mg, L-dopa 140 mg plasma samples were taken at pre-dose, 30, 60, 90 and 120 minutes post-dose. For the L-dopa 70 mg/carbidopa 7 mg treatment arm, plasma samples were taken at pre-dose, 5, 10, 15, 30, 45, 60, 90 and 120 minutes post-dose.
Time Frame: For L-dopa 35 mg, 70 mg, 140 mg plasma samples were taken at pre-dose, 30, 60, 90 and 120 minutes post-dose. For L-dopa 70 mg/carbidopa 7 mg, plasma samples were taken at pre-dose, 5, 10, 15, 30, 45, 60, 90 and 120 min
Population: Subjects who received L-dopa or L-dopa/carbidopa. Placebo subjects therefore not included.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours*ng/mL | 240.71 (117.819) | 463.49 (260.093) | 725.29 (456.566) | 552.75 (177.979)

3. Secondary Outcome: Cmax of L-dopa
Description: Maximum Observed Plasma Concentration of L-dopa from Time = 0 to Time = 2 hours post dose. For the L-dopa 35 mg, L-dopa 70 mg, L-dopa 140 mg plasma samples were taken at pre-dose, 30, 60, 90 and 120 minutes post-dose. For the L-dopa 70 mg/carbidopa 7 mg treatment arm, plasma samples were taken at pre-dose, 5, 10, 15, 30, 45, 60, 90 and 120 minutes post-dose.
Time Frame: For L-dopa 35 mg, 70 mg, 140 mg plasma samples were taken at pre-dose, 30, 60, 90 and 120 minutes post-dose. For L-dopa 70 mg/carbidopa 7 mg, plasma samples were taken at pre-dose, 5, 10, 15, 30, 45, 60, 90 and 120 minutes post-dose.
Population: Subjects who received L-dopa. Placebo subjects not included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 185.80 (78.144) | 362.68 (195.265) | 643.65 (462.469) | 445.75 (183.746)

4. Secondary Outcome: Tmax of L-dopa
Description: Time to Reach the Maximum Plasma Concentration (Cmax) of L-dopa
Time Frame: as for outcome 3
Population: Subjects who received L-dopa. Placebo subjects not included.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
minutes | 60.17 (37.950) | 66.00 (38.735) | 70.00 (15.505) | 92.00 (27.481)

5. Secondary Outcome: Mean Change From Baseline in MDS-UPDRS Score Over 2 Hours for C1, C2, C3 and Change From Baseline at 30, 60, 90, 120 Minutes for C4, in MDS-UPDRS Part III Score
Description: MDS-UPDRS is a clinimetric assessment of subjective and objective symptoms and signs of Parkinson's disease created by the Movement Disorder Society with high internal consistency. MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The subscale used in this study is Part III, motor examination (18 items). The subscale has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. Maximum score is 132, minimum is zero. High score means worse outcome. For the L-dopa 35 mg, L-dopa 70 mg, L-dopa 140 mg treatment groups, assessment occurred at pre-dose, 15, 30, 45, 60, 90 and 120 minutes post-dose. For the L-dopa 70 mg/carbidopa 7 mg treatment arm, assessment occurred at pre-dose, 30, 60, 90 and 120 minutes post-dose.
Time Frame: For L-dopa 35 mg, 70 mg, 140 mg, assessment occurred at pre-dose, 15, 30, 45, 60, 90 and 120 minutes post-dose. For L-dopa 70 mg/carbidopa 7 mg, assessment occurred at pre-dose, 30, 60, 90 and 120 minutes post-dose.
Population: All participants were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
score on a scale
  15 minutes: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  15 minutes | -3.5 (3.89) | -4.5 (4.46) | 0.8 (9.20) | -9.0 (6.16) | NA (NA) — Participants in this arm were not tested at this time point.
  30 minutes | -8.5 (6.52) | -6.7 (4.89) | -8.5 (9.09) | -12.7 (7.79) | -3.7 (3.83)
  45 minutes: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  45 minutes | -13.5 (7.09) | -4.7 (4.03) | -12.8 (11.05) | -13.7 (8.91) | NA (NA) — Participants in this arm were not tested at this time point.
  60 minutes | -12.5 (7.87) | -6.8 (4.54) | -15.7 (9.58) | -13.5 (8.29) | -0.8 (10.63)
  90 minutes | -10.8 (9.35) | -10.3 (13.56) | -15.5 (10.03) | -9.0 (5.76) | -3.7 (10.76)
  120 minutes | -8.8 (10.61) | -11.0 (9.47) | -13.8 (11.97) | -7.2 (9.09) | -3.2 (9.22)

6. Secondary Outcome: Time to Response (Defined as Improvement of 30% in MDS-UPDRS Part III Score From Baseline)
Description: MDS-UPDRS is a clinimetric assessment of subjective and objective symptoms and signs of Parkinson's disease created by the Movement Disorder Society with high internal consistency. MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The subscale used in this study is Part III, motor examination (18 items). The subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: 2 hours
Population: All participants were analyzed.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
minutes | 45.0 [35.0 to NA] — The upper bound of the 95% CI could not be calculated due to the number of participants not achieving a response in the analysis time frame | NA [40.0 to NA] — The median and the upper bound of the 95% CI could not be calculated due to the number of participants not achieving a response in the analysis time frame | 54.0 [15.0 to NA] — The upper bound of the 95% CI could not be calculated due to the number of participants not achieving a response in the analysis time frame | 30.0 [15.0 to NA] — The upper bound of the 95% CI could not be calculated due to the number of participants not achieving a response in the analysis time frame | NA [32.0 to NA] — The median and the upper bound of the 95% CI could not be calculated due to the number of participants not achieving a response in the analysis time frame

7. Secondary Outcome: Cumulative Number of Responders (Defined as Improvement of 30% in MDS-UPDRS Part III Score From Baseline)
Description: as for outcome 6
Time Frame: From time = 0 to 2 hours post-dose
Population: All participants were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participants
  15 minutes: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  15 minutes | 0 | 0 | 1 | 2 | NA — Subjects in this arm were not analyzed at this time point.
  30 minutes | 3 | 1 | 1 | 5 | 1
  45 minutes: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  45 minutes | 4 | 1 | 3 | 5 | NA — Subjects in this arm were not analyzed at this time point.
  60 minutes | 6 | 1 | 4 | 5 | 2
  90 minutes | 6 | 2 | 5 | 5 | 3
  120 minutes | 6 | 2 | 5 | 5 | 3

8. Secondary Outcome: Area Under the Curve (AUC) of Change From Baseline in MDS-UPDRS Part III Scores
Description: as for outcome 6
Time Frame: For L-dopa 35 mg, 70 mg, 140 mg, assessments were made at pre-dose, 15, 30, 45, 60, 90, 120 minutes post-dose. For L-dopa 70 mg/carbidopa 7 mg, assessments were made at pre-dose, 50, 60, 90, 120 minutes post-dose.
Population: All participants were included in the analysis
Measure: Mean (Standard Deviation); unit: change in score*minutes
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
change in score*minutes
  15 minutes: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  15 minutes | -26.25 (29.144) | -33.50 (33.697) | 7.00 (69.206) | -67.50 (46.233) | NA (NA) — Participants in this arm were not assessed at this time point.
  30 minutes | -237.63 (276.197) | -138.58 (138.105) | -50.50 (203.053) | -232.83 (153.638) | -230.08 (250.832)
  45 minutes: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  45 minutes | -264.92 (178.969) | -201.92 (162.256) | -210.50 (334.216) | -426.83 (274.566) | NA (NA) — Participants in this arm were not assessed at this time point.
  60 minutes | -573.88 (371.782) | -296.50 (241.271) | -424.25 (464.545) | -630.58 (401.947) | -295.25 (412.042)
  90 minutes | -919.75 (530.872) | -575.17 (486.241) | -896.67 (671.116) | -968.08 (587.629) | -362.75 (676.456)
  120 minutes | -1215.75 (765.287) | -903.67 (804.196) | -1324.83 (863.122) | -1210.58 (714.512) | -465.25 (932.842)

9. Secondary Outcome: Mean Maximum Change From Baseline in MDS-UPDRS Part III Score
Description: MDS-UPDRS is a clinimetric assessment of subjective and objective symptoms and signs of Parkinson's disease created by the Movement Disorder Society with high internal consistency. MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The subscale used in this study is Part III, motor examination (18 items). The subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The total of the subscales has a maximum value of 132 and a minimum value of zero. Lower scores indicate better motor function. A negative change from baseline indicates improved motor function.
Time Frame: From time = 0 to 2 hours post-dose
Population: All subjects were included in this analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
score on a scale | -15.5 (6.35) | -14.0 (11.15) | -20.3 (11.18) | -15.3 (8.12) | -7.5 (6.72)

10. Secondary Outcome: Subjective Time to "ON" as Evaluated by the Investigator
Description: Investigators will evaluate subjects' fluctuations in motor functions at 15, 30, 45, 60, 90, 120, and 240 minutes post-dose to determine if they are "ON".
Time Frame: 4 hours
Population: All participants were included in the analysis
Measure: Median (Full Range); unit: minutes
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
minutes | 45.0 [30 to 240] | 240.0 [90 to NA] — One or more subjects in this arm did not achieve ON by the end of the assessment period. Therefore upper range was >240 minutes. | 30.0 [15 to 240] | 30.0 [15 to 240] | 240.0 [30 to 240]

11. Secondary Outcome: Assessment of Time to "ON" as Evaluated by Subject Self-assessment
Description: Subjects were asked to provide self-assessments at 15, 30, 45, 60, 90, 120, and 240 minutes post-dose as to whether they considered themselves to be "ON".
Time Frame: 4 hours
Population: All participants were included in the analysis.
Measure: Median (Full Range); unit: minutes
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
minutes | 40.0 [15 to 240] | 240.0 [95 to NA] — One or more participants in this arm did not perceive themselves to be "ON" by the end of the assessment period, therefore the full range is 95 to >240 minutes | 39.0 [15 to 240] | 30.0 [15 to 240] | 232.5 [31 to 240]

12. Secondary Outcome: AUC0-2h for Carbidopa
Description: Area under the concentration time curve for carbidopa
Time Frame: Plasma samples were taken at pre-dose, 5, 10, 15, 30, 45, 60, 90 and 120 minutes post-dose and AUC calculated from these from time 0 to 120 minutes.
Population: Subjects who received the combination of L-dopa/carbidopa
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 6
hours*ng/mL | 114.80 (30.384)

13. Secondary Outcome: Cmax of Carbidopa
Description: Maximum concentration of carbidopa
Time Frame: For L-dopa 70 mg/carbidopa 7 mg, plasma samples were taken at pre-dose, 5, 10, 15, 30, 45, 60, 90 and 120 minutes post-dose.
Population: Subjects who received L-dopa/carbidopa
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 6
ng/mL | 80.23 (22.945)

14. Secondary Outcome: Tmax of Carbidopa
Description: Time to reach the maximum concentration of carbidopa
Time Frame: as for outcome 13
Population: Subjects who received L-dopa/carbidopa
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 6
minutes | 44.50 (13.882)

15. Secondary Outcome: Duration of Response, Where Response is Defined as an Improvement of 30% in MDS-UPDRS Part III Score From Baseline.
Description: MDS-UPDRS is a clinimetric assessment of subjective and objective symptoms and signs of Parkinson's disease created by the Movement Disorder Society with high internal consistency. MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The subscale used in this study is Part III, motor examination (18 items). The subscale has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. Maximum score is 132, minimum is zero. High score means worse outcome.
Time Frame: 2 hours
Population: All participants were analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
minutes | 66.9 (48.35) | 23.3 (36.70) | 57.3 (42.72) | 37.5 (42.25) | 15.0 (25.10)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Placebo | L-dopa 35 mg | L-dopa 70 mg | L-dopa 140 mg | L-dopa 70 mg/Carbidopa 7 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/8 | 5/6 | 3/6 | 4/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | L-dopa 35 mg (N=6) | L-dopa 70 mg (N=6) | L-dopa 140 mg (N=6) | L-dopa 70 mg/Carbidopa 7 mg (N=6)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
paranasal sinus hyposecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03541356/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT03541356/SAP_001.pdf